CLINICAL TRIAL: NCT06846463
Title: Phase 2 Trial Utilizing Zanubrutinib in Patients With Diffuse Large B-cell Lymphoma and MYD88 L265P Mutations, CD79B Mutations, NOTCH1 Truncation or Who Are CD5+ by IHC.
Brief Title: Zanubrutinib in Patients With DLBCL and MYD88 or NOTCH1 Mutation or CD5+
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-24-21151; HM20031622 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B-cell Lymphoma; DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Agent Administration (Experimental): Zanubrutinib is administered as capsules for oral intake at one of the following dosages based on the discretion of the treating physician:
  * 160 mg (two 80-mg capsules) twice daily
  * 320 mg (four 80-mg capsules) once daily
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Investigational Agent Administration. Zanubrutinib will be first administered on Cycle 2 Day 1 of rituximab, cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), vincristine sulfate (Oncovin), and prednisone (R-CHOP). It is up to the discretion of the treating physician how many cycles of R-CHOP the treatment would require, but it is not to exceed 6 cycles of R-CHOP and 5 cycles of zanubrutinib. The number of cycles of R-CHOP should be per standard of care, with the number of zanubrutinib cycles being 1 less than the number of total R-CHOP cycles.

SUMMARY:
This study is a single-arm, open label, non-randomized, phase 2 trial of zanubrutinib in patients with diffuse large B-cell lymphoma (DLBCL) who have an MYD88 L265P mutation, a CD79B mutation, a NOTCH1 truncation, or who are CD5+ by immunohistochemistry (IHC).

DETAILED DESCRIPTION:
The purpose of this study is to compare effects of adding zanubrutinib to the usual chemotherapy in patients with diffuse large B-cell lymphoma (DLBCL) who have an MYD88 L265P mutation, a CD79B mutation, a NOTCH1 truncation, or who are CD5+ by IHC. In those patients with mutations or IHC result, we propose treating with zanubrutinib plus rituximab, cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), vincristine sulfate (Oncovin), and prednisone (R-CHOP). Patients will be monitored with standard imaging; minimal residual disease (MRD) testing will be optional. The primary outcome is the complete response rate. The secondary outcome is EFS at 2 years. When available, MRD studies will be correlated to response. Patients with aggressive B-cell lymphoma with MYC and BCL-2 and/or BCL-6 mutations will be excluded, as will patients with HIV. Zanubrutinib will be first administered on Cycle 2 Day 1 of R-CHOP. It is up to the discretion of the treating physician how many cycles of R-CHOP the treatment would require, but it is not to exceed 6 cycles of R-CHOP and 5 cycles of zanubrutinib. The number of cycles of R-CHOP should be per standard of care, with the number of zanubrutinib cycles being 1 less than the number of total R-CHOP cycles. Patients will be followed up every 3 months for 24 months after removal from protocol therapy or until death, whichever occurs first. There will be an extended follow-up period of up to 5 years from end of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a documented pathologic diagnosis of DLBCL at any stage.
* Must have documented MYD88 L265P, CD79B, or NOTCH1 truncation mutation or be CD5+ by IHC.
* Age ≥18 years on the day of signing the informed consent form.
* Patients must have measurable disease on Positron Emission Tomography-Computed Tomography scan (CT/PET) imaging.
* Patient must have received no more than one cycle of R-CHOP prior to enrollment. Length of time between first R-CHOP treatment and planned 2nd R-CHOP treatment should vary by no more than 21 days ± 3 days.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Adequate bone marrow function as defined by:

  * Absolute neutrophil count (ANC) ≥1000/mm3, except for patients with bone marrow involvement in which ANC must be ≥500/mm3.
  * Platelet ≥75,000/mm3, except for patients with bone marrow involvement in which the platelet count must be ≥30,000/mm3.
  * Hemoglobin ≥7 g/dL, after transfusion if necessary
* Adequate organ function defined as:

  * Creatinine clearance ≥30 mL/min as estimated by the Cockcroft-Gault equation.
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase, and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase ≤2.5 × upper limit of normal (ULN).
  * Serum total bilirubin ≤3 x ULN (except patients with Gilberts syndrome 3g/dl).
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use one of the following highly effective forms of birth control during the treatment and for 1 month following completion of study treatment for women and for 1 week following completion of study treatment for men.

  * combined (estrogen and progestogen containing) hormonal contraception:
* oral
* intravaginal
* transdermal

  * progestogen-only hormonal contraception associated with inhibition of ovulation
* oral
* injectable
* implantable

  * intrauterine device (IUD)
  * intrauterine hormone-releasing system (IUS)
  * bilateral tubal occlusion
  * vasectomized partner
  * heterosexual abstinence
* Patients must not have any known allergies, hypersensitivity or intolerance to corticosteroids or monoclonal antibodies.
* Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments.

Exclusion Criteria:

* Patients with high grade B-cell lymphoma with myelocytomatosis oncogene /immunoglobulin heavy-chain (MYC)/IGH and BCL-2 rearrangements.
* Patients with brain metastasis.
* Patients with peripheral neuropathy CTCAE grade ≥2.
* Any uncontrolled or clinically significant cardiovascular disease including the following:

  * Myocardial infarction within 6 months before screening.
  * Unstable angina within 3 months before screening.
  * New York Heart Association class III or IV congestive heart failure.
  * History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes).
* Prior malignancy within the past 3 years, except for curatively treated basal or squamous cell skin cancer, non-muscle-invasive bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 prostate cancer.
* History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention.
* History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.
* Severe or debilitating pulmonary disease in the opinion of the treating investigator.
* Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Active fungal, bacterial and/or viral infection requiring systemic therapy.
* Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs.
* Active infection with HIV, or serologic status reflecting active hepatitis B or C infection as follows:

  * Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) DNA is undetectable (< 20 IU), and if they are willing to undergo monitoring every 4 weeks for HBV reactivation.
  * Presence of hepatitis C virus (HCV) antibody. Patients with presence of HCV antibody are eligible if HCV RNA is undetectable.
* Major surgery within 4 weeks of the first dose of study drug.
* Pregnant or lactating women.
* Left ventricular ejection fraction (LVEF) <55% on screening echocardiogram.
* Vaccination or requirement for vaccination with a live vaccine within 28 days prior to the first dose of study drug or at any time during planned study treatment.
* Hypersensitivity to zanubrutinib, rituximab, cyclophosphamide, doxorubicin, vincristine, or prednisone.
* Requires ongoing treatment with a strong CYP3A inducer (Table 3).
* Concurrent participation in another therapeutic clinical trial.
* Active and/or ongoing autoimmune anemia and/or autoimmune thrombocytopenia (eg, idiopathic thrombocytopenia purpura).
* Requires ongoing treatment with warfarin or warfarin derivatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Assess efficacy of adding oral zanubrutinib to R-CHOP in patients with DLBCL who have an MYD88 L265P mutation, a CD79B mutation, a NOTCH1 truncation, or who are CD5+ by Immunohistochemistry (IHC) in achieving complete response defined by Lugano criteria | Completion of treatment through 2 years +/- 2 weeks
  Percentage of participants with complete response by immunohistochemistry (IHC).

SECONDARY OUTCOMES:
Assess efficacy of adding oral zanubrutinib in addition to R-CHOP in patients with DLBCL who have an MYD88 L265P mutation, a CD79B mutation, a NOTCH1 truncation, or who are CD5+ by IHC in achieving radiographic 2-year EFS and duration of response (DOR) | Up to 5 years following end of treatment
  Percentage of participants with Radiographic 2-year event free survival (EFS) as defined by the time after the first treatment until the date of first treatment failure or death.
Assess the safety of adding oral zanubrutinib in addition to R-CHOP in patients with DLBCL who have a MYD88 L265P mutation, a CD79B mutation, a NOTCH1 truncation, or who are CD5+ by IHC by observing adverse events (AE's) of special interest. | Baseline, during protocol treatment, though 2 year follow-up
  Occurrence of hematologic and non-hematologic toxicity as defined by the percent of patients who have each toxicity over all 6 cycles. Adverse events of special interest hematologic toxicity including:
  * Neutropenic fever
  * All grades of anemia
  * Neutropenia and thrombocytopenia as defined by the percent of patients who have this AE over all 6 cycles.
  Non-hematologic toxicity including:
  * Fungal infection
  * Bacterial pneumonia
  * Rash as defined by the percent of patients who have this AE over all 6 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Hough, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD at this time.